CLINICAL TRIAL: NCT06316193
Title: The Use of the Diary in Neonatal Pathology: a Mixed-method Study for Collecting and Analyzing the Experience of Parents and Health Care Personnel.
Acronym: DiaPaNeo
Status: Recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Roberta Ranzani, Nurse, Principal Investigator, IRCCS Ospedale San Raffaele
Other Study IDs: DiaPaNeo
Record Dates: First submitted 2024-03-02; First posted 2024-03-18 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Experience, Life; Stress; Depression, Postpartum; Support, Family
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diary — The diary is the tool through which the experiences and experiences of the parents of infants admitted to Neonatal Pathology and included in the study and the health care personnel who decide to participate will be collected and analyzed. This tool is given to the parents of infants included in the study in the first few days of the infant's stay (by the third day after admission), subject to the parents' written consent, accompanied by a brief letter of introduction to the diary itself, written by the nurses on the ward. This tool has been part of current clinical practice since January 2023.

SUMMARY:
The study is mixed-methods (qualitative + quantitative observational cross-sectional) and the aims are to explore the use of diaries by parents of newborns admitted to Neonatal Pathology and to describe some variables related to their experience during their children's hospitalization, such as: stress level, postpartum depression and perceived support. The diary that will be analyzed is already part of current clinical practice. Study population:

* Parents of premature infants with gestational age less than or equal to 35 weeks and infants with birth weight less than or equal to 2kg admitted to Neonatal Pathology of San Raffaele Hospital.
* Health workers of the O.U. of Neonatal Pathology.

ELIGIBILITY:
Inclusion Criteria:

for the parents:

* signed informed consent;
* parents of premature infant with gestational age less than or equal to 35 gestational weeks and with birth weight less than or equal to 2kg.

for healthcare providers:

* healthcare personnel from the O.U. of Neonatal Pathology;
* signed informed consent.

Exclusion Criteria:

for parents:

* non-understanding or inability to express themselves in Italian language;
* parent of premature infant with gestational age greater than 35 gestational weeks and with birth weight greater than 2kg
* unsigned informed consent.

for health workers:

* healthcare personnel not working in the O.U. of Neonatal Pathology;
* unsigned informed consen

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants are parents of premature infants with gestational age less than or equal to 35 weeks and infants with birth weight less than or equal to 2kg admitted to Neonatal Pathology of San Raffaele Hospital, and health workers of the O.U. of Neonatal Pathology.
  For both the qualitative and quantitative studies, it is planned to enroll at least 15 infants and their parents; at least 10 health workers who participated in the diary compilation. The study is monocentric, only the U.O. of Neonatal Pathology is involved in the study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
The objective of the qualitative phase is to provide a description of the experience of the parents of infants admitted to Neonatal Pathology and the healthcare personnel who participated in the compilation of the diary. | Data collection will take place between April 15, 2024 and April 15, 2025.
  The diary is the tool through which the experiences of the parents of infants and included in the study and the healthcare personnel who decide to participate will be collected and analyzed. It is given to the parents in the first few days of the infant's stay, subject to the parents' written consent, accompanied by a brief letter of introduction to the diary itself, written by the nurses on the ward. This tool has been part of current clinical practice since January 2023.The diary consists of an A5-sized notebook with ruled sheets. The pages of the diary are blank, with no rigid structure,so that the parents are free to write his or her own thoughts.

SECONDARY OUTCOMES:
The quantitative phase includes as data collection tools a set of instruments validated in the Italian context and selected in relation to the variables to be measured. The instruments will be administered by one of the appropriately trained nurses. | Data collection will take place between April 15, 2024 and April 15, 2025.
  The quantitative phase includes as data collection tools:
  * socio-demographic profile of the parents: for both parents, data will be collected on year of birth, gender, nationality, education level, occupation, family status, presence of other children, similar lived experiences, support from other figures close to the family (e.g., grandparents), distance from the hospital (km), religion, taking care of by a psychologist, previous experience of hospitalization in Neonatal Pathology. For the mother only: obstetric history;
  * socio-demographic profile of the newborn: gestational age, birth weight, twins, other pathologies present, type of delivery, Apgar score and prenatal diagnosis;
  * socio-demographic profile of the healthcare workers: year of birth, gender, occupational qualification, educational qualification, years of service in general and years of service in Neonatal Pathology.
The quantitative phase includes as data collection tools a set of instruments validated in the Italian context and selected in relation to the variables to be measured. Stressor Scale (PSS). | Data collection will take place between April 15, 2024 and April 15, 2025.
  Parental stress is a form of stress characterized by adverse psychological and physiological reactions resulting from attempts to adapt to the demands of parenting. This variable will be assessed in both parents with the PSS. The scale consists of 26 items that assess three dimensions related to parents' stress during their children's stay in the NICU:
  * lights and sounds (6 items): stress related to the physical environment of the NICU;
  * infant behavior and appearance (13 items): stress related to infant appearance and behavior;
  * parental role alteration (7 items): stress related to the alteration of the expected parental role.
  Parents are asked to rate each item with a score ranging from 1 to 5, to indicate how stressful the situation described by each item was for them (1 not at all stressful - 5 extremely stressful, NA not applicable if the experience was not experienced).The higher the score obtained by summing the scores attributed to the individual items, the higher the
The quantitative phase includes as data collection tools a set of instruments validated in the Italian context and selected in relation to the variables to be measured. Edinburgh Postnatal Depression Scale (EPDS). | Data collection will take place between April 15, 2024 and April 15, 2025.
  Postpartum depression is one of the most common complications following childbirth. Postpartum depression also has negative effects on the child's behavioral, emotional and cognitive development. Symptoms of such depression include: mood lability, anxiety, irritability, feelings of overwhelm and obsessive worries or concerns, often related to the health, nutrition and safety of the baby. This variable will be collected only in mothers with the Edinburgh Postnatal Depression Scale (EPDS). This instrument is a self-assessment scale for detecting the onset of postpartum depression. It consists of 10 items answered on a 4-point Likert scale (0 - 3). In case the score obtained is higher than 12, the risk of postpartum depression should not be neglected and a specialist should be consulted. The tool has been validated in the Italian context. It will be administered only to mothers.
The quantitative phase includes as data collection tools a set of instruments validated in the Italian context and selected in relation to the variables to be measured. The Nurse Parental Support Tool (NPST). | Data collection will take place between April 15, 2024 and April 15, 2025.
  Parents' perceived support from medical/nursing staff: a successful relationship between parents and the care team includes parents' exchange of information, trust, and education about their children. Optimal parental caretaking by health care staff significantly reduces parental stress. The variable will be measured with The Nurse Parental Support Tool (NPST). This scale assesses parents' perceptions of their caregiving by the medical/nursing staff; it asks parents' perceptions, making explicit how often the health care staff helped them during their child's hospitalization. The scale consists of 21 items, multiple-choice, scored from 1 to 5 (1 almost never - 5 almost always). Adding up the scores for each item, higher scores reflect better parental assignment taken by the medical/nursing staff. The instrument has been validated in the Italian context

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No